CLINICAL TRIAL: NCT07303257
Title: Quality of Life After Glaucoma Surgery: Evaluating the Patient Perspective Across Surgical Options - G-SCOPE (Glaucoma Surgery - Comparative Patient Evaluation)
Brief Title: Quality of Life After Glaucoma Surgery: Evaluating the Patient Perspective Across Surgical Options
Acronym: G-SCOPE
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL25_0896; 2025-A02669-40 (Other: ANSM)
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Glaucoma Eye; Open-angle Glaucoma; Closed-Angle Glaucoma; Pseudo Exfoliative Syndrome; Pigmentary Glaucoma
Keywords: Glaucoma; Trabeculectomy; Sclerectomy; PreserFlo® Micro Shunt; Quality of life; Glaucome Surgery; MIGS; NEI-VFQ 25 (National Eye Institute- Visual Function Questionnaire 25)
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma, Angle-Closure; Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult with open-angle/angle-closure or exfoliative or pigmentary glaucoma and a surgical indication: Adult patient with different stage of glaucoma and a surgical indication for sclerectomy + Mitomycin, PRESERFLO + Mitomycin, or trabeculectomy + Mitomycin.
  .
  Interventions: Other: NEI-VFQ-25 (National Eye Institute Visual Function Questionnaire-25).

INTERVENTIONS:
Other: NEI-VFQ-25 (National Eye Institute Visual Function Questionnaire-25). — The NEI-VFQ-25 questionnaire, translated into French and validated by the French National Authority for Health (HAS), is used to assess quality of life related to visual function.
  This questionnaire includes 25 items divided into 11 subdomains assessing vision-related functioning and 1 subdomain assessing general health status (see appendix for the detailed list).
  The composite score ranges from 0 to 100, with lower scores indicating a poorer perceived level of health and visual functioning.

SUMMARY:
Glaucoma surgery currently relies on a wide therapeutic arsenal, ranging from conventional filtering surgeries to minimally invasive glaucoma surgery (MIGS). These techniques offer distinct efficacy and safety profiles, allowing tailored management across a broad spectrum of patients. Traditionally, surgical success has been evaluated using objective clinical outcomes, such as intraocular pressure (IOP) reduction and decreased reliance on topical treatments.

However, the shift toward patient-centered medicine now requires consideration of the patient's perspective, including their subjective experience and the impact of treatment on quality of life. In this context, quality-of-life assessment has become a key component, promoting therapeutic alliance and patient adherence to care pathways. Despite its importance, few studies have evaluated and compared quality of life after glaucoma surgery using comparable surgical techniques.

Furthermore, to our knowledge, no study has specifically assessed the independent effect of postoperative follow-up on quality of life after filtering surgery with a bleb. Given that postoperative management can be prolonged and demanding, it may significantly influence patients' perceptions of surgical outcomes and overall well-being.

This study aims to address these gaps by providing a more comprehensive evaluation of the impact of glaucoma surgery beyond traditional clinical outcomes. It may represent a first step toward the development of a more appropriate assessment tool that incorporates the realities of postoperative follow-up and the specific experiences of patients undergoing filtering surgery.

The study is based on the following hypotheses: filtering glaucoma surgery preserves patients' quality of life, with a stable NEI VFQ-25 score at six months postoperatively; postoperative quality of life may be influenced by the patient's postoperative care pathway; and quality-of-life scores remain correlated with objective clinical parameters, including intraocular pressure, visual acuity, medical treatment burden, and visual field damage.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years with an indication for glaucoma surgical treatment
* Eligible surgical procedures: Preserflo™ MicroShunt with mitomycin C, Trabeculectomy with mitomycin C or non-penetrating deep sclerectomy with mitomycin C
* Unilateral or bilateral glaucoma, open-angle or angle-closure, at early, moderate, or advanced stages
* Pseudoxexfoliative or pigmentary glaucoma
* Secondary glaucoma, including: uveitic glaucoma, Steroid-induced glaucoma, traumatic glaucoma
* Written informed consent obtained prior to study participation

Exclusion Criteria:

* Congenital glaucoma
* Refractory glaucoma with a history of multiple previous surgeries
* Ophthalmologic surgery within 6 months prior to inclusion
* Severe visual co-morbidities (age-related macular degeneration, severe diabetic retinopathy, retinal degeneration, or similar conditions)
* Expected difficulty with follow-up including poor anticipated compliance, planned travel or prolonged absence during the follow-up period
* Illiteracy, inability to speak French or impaired cognitive capacity preventing adequate understanding of the study
* Patients with a significant pre-existing impairment in quality of life attributable to a progressive physical illness or a neuropsychiatric disorder.
* Patients under curatorship or guardianship
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glaucoma patients aged ≥ 18 years, operated on using one of the following 3 types of surgery: Trabeculectomy , Deep non-perforating sclerectomy or Preserflo
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Quality of life score from the NEI-VFQ-25 (National Eye Institute Visual Function Questionnaire-25). | Pre-operative period and 6 months after intervention
  To evaluate, in adult patients undergoing glaucoma surgery, the change in NEI-VFQ 25 quality of life score between the pre-operative period and 6ᵉ months post-operatively, regardless of the surgical technique used.

SECONDARY OUTCOMES:
Comparison of NEI-VFQ-25 scores between surgical techniques | 6 months postoperatively (M6)
  Comparison of postoperative vision-related quality-of-life outcomes across the different glaucoma surgical techniques, assessed using the global NEI-VFQ-25 score at 6 months after surgery.
  The questionnaire yields a total score ranging from 0 to 100, with higher scores corresponding to a positive outcome.
  It will be self-completed by the patient, with an estimated completion time of approximately 15 minutes. No changes will be made to the department's standard postoperative follow-up protocol.
Correlation between NEI-VFQ-25 score and postoperative clinical parameters | Postoperative visits at Month 3 (M3)
  To assess the relationship between vision-related quality-of-life outcomes, measured by the NEI-VFQ-25 score, and objective postoperative clinical results.
Correlation between NEI-VFQ-25 score and postoperative clinical parameters | Postoperative visits at Month 6 (M6)
  To assess the relationship between vision-related quality-of-life outcomes, measured by the NEI-VFQ-25 score, and objective postoperative clinical results.
Impact of postoperative follow-up on NEI-VFQ-25 quality-of-life scores at 3 months | Prospective collection of postoperative follow-up data through Month 3 (M3)
  To evaluate the effect of postoperative management-including adjunctive procedures, number of follow-up visits, and the occurrence of complications-on the NEI-VFQ-25 quality-of-life score in patients undergoing glaucoma surgery with a filtering bleb.
Impact of postoperative follow-up on NEI-VFQ-25 quality-of-life scores at 6 months | Prospective collection of postoperative follow-up data through Month 6 (M6)
  To evaluate the effect of postoperative management-including adjunctive procedures, number of follow-up visits, and the occurrence of complications-on the NEI-VFQ-25 quality-of-life score in patients undergoing glaucoma surgery with a filtering bleb.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Ophtalmologie, Hôpital de La Croix Rousse, Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No